CLINICAL TRIAL: NCT00859573
Title: Clinical Efficacy of Modafinil in Recently-Abstinent Methamphetamine-Dependent Volunteers
Brief Title: Modafinil for Methamphetamine Dependence
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to lack of funding.
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P50 DA018197-104386; P50DA018197 (NIH)
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Results first posted 2011-07-15 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-10

CONDITIONS: Methamphetamine Dependence
MeSH Terms: interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. Modafinil (Active Comparator)
  Interventions: Drug: Modafinil
- 2: Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Modafinil — 400 mg/day
  Arms: 1. Modafinil
Drug: Placebo — inactive substance
  Arms: 2: Placebo

SUMMARY:
Fifty methamphetamine dependent treatment-seeking volunteers will be enrolled in this 10 week, double bind, placebo controlled, randomized clinical trial to receive either modafinil or placebo. Eligible subjects will reside at the Recovery Centers of Arkansas residential facility to achieve initial abstinence and be inducted onto study medication during wks 1-2. Then during wks 3-10, subjects participate on an outpatient basis, receiving weekly psychotherapy while continuing to receive study medications. Urine samples will be collected thrice weekly and self reports weekly to assess methamphetamine use. It is hoped that the results of this study will contribute to our understanding of which types of agents may be good candidates for further development as potential treatment agents for this disorder.

ELIGIBILITY:
Inclusion Criteria:

18-65 years old. For the neurophysiological measures portion of the study subjects will be included if they are between the ages of 20-65 because the P50 potential is not fully developed in children and adolescents (Rasco 2000).

* not currently enrolled in a treatment program
* subjects must have a history of methamphetamine use with recent use confirmed by a positive urine toxicology screen for amphetamines during the month prior to study entry
* subjects must meet DSM-IV criteria for amphetamine dependence as assessed by the substance abuse section of the Structured Clinical Interview for DSM-IV (SCID)
* women of childbearing age must have a negative pregnancy test to enroll in this study, agree to monthly pregnancy testing, and agree to use appropriate forms of birth control for the duration of the study.

Exclusion Criteria:

* current diagnosis of alcohol, opiate, or sedative physical dependence
* ill health (e.g., major cardiovascular, renal, endocrine, hepatic disorder)
* history of schizophrenia, or bipolar type I disorder
* present or recent use of over-the-counter or prescription psychoactive drug or drug(s) that would be expected to have major interaction with drug to be tested
* medical contraindication to receiving study medications (e.g., allergy to modafinil, treatment with cyclosporine, clomipramine or desipramine)
* current suicidality or psychosis
* Liver function tests (i.e., liver enzymes) greater than three times normal levels
* pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-04; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mancino, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 20 participants were recruited into the study between 5/26/2009 and 3/30/2010. However, only 9 participants entered the study with 11 dropping out during the consent or intake process. They were recruited from newspaper advertisements and word-of-mouth advertising and who meet the following criteria.
Groups:
- Modafinil: Modafinil 400mg orally once daily
- Placebo: Two placebo tablets orally once daily
Period: Overall Study
Arm/Group | Modafinil | Placebo
Started | 6 | 3
Completed | 1 | 1
Not Completed | 5 | 2
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Modafinil | Placebo | Total
Number analyzed (Participants) | 6 | 3 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 9
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.25 (2.87) | 35.88 (12.15) | 32.56 (9.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Mean Treatment Effectiveness Scores
Description: Number of negative drug screens for methamphetamine during the study (every negative drug screen obtained is counted as 1 negative drug screen)divided by the total possible number of drug screens during the 6 week post residential phase of trial(participants provided 3 drug screens per week so the expected number of drug screens total is 18.This does include week 8. Missing drug screens are counted as positive.# negative drug screens/18. Minimum score is 0 and maximum score is 1. The higher the score the better the outcome. The mean of the individual treatment effectiveness scores is reported.
Time Frame: thrice weekly from week 3 through week 8
Population: Participants that completed the 2 week residential treatment and entered the outpatient phase with intent to treat and missing urines treated as positive urines.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Placebo: Participants received 2 capsules placebo orally daily
- Modafinil: Modafinil 400mg orally daily
Arm/Group | Placebo | Modafinil
Number analyzed (Participants) | 2 | 3
scores on a scale | 0.5625 (0.38) | .333 (.31)

ADVERSE EVENTS:
Arm/Group | Modafinil | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3
Other Adverse Events (participants affected / at risk) | 4/6 | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Modafinil (N=6) | Placebo (N=3)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Weight loss (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed. Small number of completers leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes